CLINICAL TRIAL: NCT03357744
Title: Face-to-face Interviews or Written Self-report Questionnaires: The Distress-barometer as a Screening Instrument for Psychosocial Complaints in Patients With Breast Cancer
Brief Title: The Distress-barometer: Face-to-face Interviews or Written Self-report Questionnaires?
Status: Completed | Type: Observational
Sponsor: KU Leuven (Other)
Collaborators: Ziekenhuis Oost-Limburg (Other)
Responsible Party: Principal Investigator, Bert Aertgeerts, Prof. Dr., KU Leuven
Other Study IDs: Katholieke Universiteit Leuven
Record Dates: First submitted 2017-11-22; First posted 2017-11-30 (Actual); Last update posted 2017-11-30 (Actual); Status verified 2017-11

CONDITIONS: Breast Cancer
Keywords: distress; assessment methods
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 2 Weeks
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: distress barometer — not applicable, observational study

SUMMARY:
Breast cancer is the most prevalent cancer among women worldwide [1]. 5 years after diagnosis, up to 87% survives. A substantial group of these survivors report reduced physical, psycho social and cognitive functioning. Therefore, it is increasingly important to screen for distress, both during and after treatment. The Distress Barometer (DB) is a valid, short screening instrument, used to detect elevated levels of distress in patients with cancer. It can be used either in a self-report questionnaire or in an interview format.

Although the DB is used in different ways, it remains unclear whether both assessment methods would generate similar results, and which format is most suitable to represent the actual level of distress. Existing literature on the DB lacks a systematic description of the relationship between the method of assessment and the patients' responses. This study questions whether the written and interview variants of the DB reveal different results in the same patients with breast cancer.

DETAILED DESCRIPTION:
Objective:

This study questions whether the written and interview variants of the DB reveal different results in the same patients with breast cancer.

Participants:

Participants were female breast cancer patients who received their diagnosis about three years before the study. Thirty patients received follow-up care in Ziekenhuis Oost-Limburg (ZOL). An additional twenty-nine patients were included in the KLIMOP-study and recruited in three Belgian hospitals (ZOL, University Hospital Leuven, Jessa Ziekenhuis). Patients were included through either clinical practice or the KLIMOP-study. All participating patients had to be able to read and understand Dutch and signed informed consent. In total, 59 patients took part in the study.

Data collection:

Two weeks after the face-to-face interview, patients with breast cancer will be provided with a written version of the DB questionnaire together with a prepaid envelop in order to evaluate the differences in written and oral versions of the DB.

Data management:

Data collection and data entries will be done by the PI and an assisting data manager. All patient data will be coded and anonymized. All other authors will have full access to the coded data (including statistical reports and tables) in the study and will be able to take responsibility for the integrity of the data and the accuracy of the data analysis.

Statistical analysis A chi-square test, accuracy and kappa statistic were performed to compare the dichotomized results of the DB between the interviews and questionnaires. Furthermore, paired t-tests were applied to compare the mean scores coming from interview and questionnaire for the CCS and for the DT.

Ethics:

This study is part of the ongoing KLIMOP-study and current clinical practice of ZOL. The study was added in the KLIMOP-study through an amendment to the Medical Ethics Committee S52097 / ML6279 (University Hospital Leuven) and a new study protocol was submitted to and approved by the Medical Ethics Committee of ZOL 16/050U.

ELIGIBILITY:
Inclusion Criteria:

* breast cancer, diagnosed 3 years ago

Exclusion Criteria:

* dementia
* no thorough command of Dutch

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Participants were female breast cancer patients who received their diagnosis about three years before the study.
Sampling Method: Non-Probability Sample
Enrollment: 59 (Actual)
Dates: Start 2016-06 (Actual); Primary Completion 2016-10 (Actual); Study Completion 2016-10 (Actual)

PRIMARY OUTCOMES:
Distress agreement between written and oral form of the questionnaire 'Distress Barometer'. | 2 weeks
  agreement between different assesment methods of distress barometer

CONTACTS AND LOCATIONS:
Overall Officials: Marjan van den Akker, PhD, Study Chair — KU Leuven

IPD SHARING:
Plan to Share IPD: No